CLINICAL TRIAL: NCT06177171
Title: A Phase I/Ib Study of Olaparib and ASTX727 in BRCA1/2- and HRD-mutated Tumors
Brief Title: Olaparib and ASTX727 in BRCA1/2- and Homologous Recombination Deficient (HRD)-Mutated Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pamela Munster (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Pamela Munster, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 23992; 5R01CA255613-02 (NIH); NCI-2023-10542 (Registry Identifier: NCI Clinical Trials Reporting Program)
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: BRCA1 Mutation; BRCA2 Mutation; BRCA Mutation; PALB2 Gene Mutation; Checkpoint Kinase 2 Gene Mutation; ATM Gene Mutation
Keywords: Homologous Recombination Deficiency; HRR Pathway
MeSH Terms: interventions — olaparib; decitabine and cedazuridine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1: Olaparib, ASTX727 (D1,D3)-Starting Dose (Experimental): Participants enrolled in the starting dose cohort will receive 300 mg Olaparib orally, twice a day (BID) on day 1 and day 14 for each 28-day cycle. Participants will also receive 35/100mg ASTX727 on days 1, and 3 of the 28-day cycle. Participants may continue study treatment indefinitely until disease progression unacceptable toxicity, withdrawal, or study closure; whichever comes first. If no DLTs are reported for the first 3 participants, an additional dose escalation cohort may open at the next dose level.
  Interventions: Drug: Olaparib; Drug: ASTX727
- Phase 1: Olaparib + ASTX727 (D1,D3,D5) (Experimental): If no DLTs are reported in the previous dose level, participants enrolled in this cohort will receive 300 mg olaparib orally, twice a day (BID) on day 1 and day 14 for each 28-day cycle. Participants will also receive 35/100mg ASTX727 on days 1, 3 and 5 of the 28-day cycle. Participants may continue study treatment indefinitely until disease progression unacceptable toxicity, withdrawal, or study closure; whichever comes first.
  Interventions: Drug: Olaparib; Drug: ASTX727
- Phase 1b: RP2D (Olaparib, ASTX727) - Dose Expansion (Experimental): Participants enrolled in this cohort will receive the RP2D based on the safety and efficacy profile determined in the Phase 1 cohorts. Participants will receive the RP2D dose of olaparib orally, twice a day (BID) on day 1 and day 14 for each 28-day cycle. Participants will also receive 35/100mg ASTX727 at the RP2D for the 28-day cycle. Participants may continue study treatment indefinitely until disease progression unacceptable toxicity, withdrawal, or study closure; whichever comes first.
  Interventions: Drug: Olaparib; Drug: ASTX727

INTERVENTIONS:
Drug: Olaparib — Given orally
  Other Names: LYNPARZA
Drug: ASTX727 — Given Orally
  Other Names: INQOVI; C-DEC

SUMMARY:
This is a single center, phase I/Ib clinical trial evaluating the combination of the poly adenosine diphosphate-ribose polymerase (PARP) inhibitor olaparib with the DNA methyltransferase (DNMT) inhibitor ASTX727, which is an oral formulation of decitabine with cedazuridine (a cytidine deaminase inhibitor that allows for oral administration). The study population consists of adults with advanced/metastatic solid tumor malignancies with germline or somatic mutations in the HRR pathway (i.e., BReast CAncer gene 1 (BRCA1), BReast CAncer gene 2(BRCA2), Partner And Localizer of BRCA2 (PALB2), ATM, and/or Checkpoint kinase 2 (CHEK2) mutations).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and tolerability of olaparib and ASTX7272 in patients with advanced solid tumors and germline or somatic mutations in the homologous recombination repair (HRR) pathway.

II. To determine the maximum tolerated dose (MTD) and recommended phase II dose (RP2D) for olaparib and ASTX7272 in patients with advanced solid tumors and germline or somatic mutations in the HRR pathway.

SECONDARY OBJECTIVES:

I. To evaluate the preliminary efficacy of the recommended dose level of olaparib and ASTX727 in patients with solid tumor malignancies and germline or somatic mutations in the HRR pathway.

EXPLORATORY OBJECTIVES:

I. To characterize HRD mutations in tumor samples and assess functional impact on HRR.

II. To assess cell free deoxyribonucleic acid (cfDNA) as a predictive biomarker of response and resistance.

III. To create patient-derived xenograft (PDX) and patient-derived organoid (PDO) models for sensitive and resistant tumors from patients treated with olaparib and ASTX727.

OUTLINE:

Testing for DNA repair mutations should occur prior to study consent or prior to enrollment via a Clinical Laboratory Improvement Amendments of 1988 (CLIA)-approved test. This study uses a 3+3 design. In phase 1, participants will be assigned to the starting dose. If no DLTs are found in the first cycle for the first 3 participants, an additional cohort at the next dose level will open for enrollment. In phase 1b, participants will receive the recommended phase 2 dose (RP2D). Participants will be followed for approximately 30 days after discontinuation of study treatment for safety, and every 16 weeks for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have histologically or cytologically confirmed advanced solid tumors (any solid tumor type) with:

   Phase I, Dose Escalation: Germline and/or somatic mutation* in one or more of the following genes: BRCA1, BRCA2, PALB2, ATM, and/or CHEK2.

   Phase Ib, Dose Expansion**:
   1. Expansion Cohort A (n=6): Germline mutation* (with or without accompanying somatic mutation) in one or more of the following genes: BRCA1, BRCA2, PALB2, ATM, and/or CHEK2;
   2. Expansion Cohort B (n=6): Germline and/or somatic mutation* in one or more of the following genes: BRCA1, BRCA2, PALB2, ATM, and/or CHEK2.

      * Testing for DNA repair mutations should occur prior to study consent or enrollment via a CLIA-approved test.
2. Has measurable disease per RECIST 1.1 as assessed by the investigator. Lesions situated in previously irradiated areas are considered measurable if progression has been demonstrated in such lesions.
3. Participants may have received any lines of prior therapy and is refractory or intolerant to therapy approved for their condition or unwilling to receive currently approved therapy.
4. Prior PARP inhibitors are allowed, provided the following two criteria are met:

   1. Participant has NOT required toxicity related dose reductions or dose delays during prior PARP inhibitor treatment; and
   2. Participant has NOT experienced any allergic reaction to PARP inhibitors.
5. Age >=18 years
6. Eastern Cooperative Oncology Group (ECOG) performance status <2, or Karnofsky >60%
7. Demonstrates adequate organ function as defined below:

   Adequate bone marrow function:
   1. hemoglobin >=10.0 g/dl
   2. absolute neutrophil count >=1,500/microliter (mcL)
   3. platelets >=100,000/mcL

   Adequate hepatic function:
   1. total bilirubin ≤ 1.5 x institutional upper limit normal (ULN)
   2. aspartate aminotransferase (AST)/(SGOT) <= 2.5 x institutional ULN
   3. alanine aminotransferase (ALT)/(SGPT) <= 2.5 x institutional ULN
   4. creatinine <= 1.5 x institutional ULN or creatinine clearance Glomerular filtration rate (GFR) >= 50 mL/min/1.73 m^2, calculated using the Cockcroft-Gault equation.
8. Ability to understand and the willingness to sign a written informed consent document.
9. Human immunodeficiency virus (HIV)-infected individuals on effective antiretroviral therapy with undetectable viral load within 6 months are eligible for this trial.
10. For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
11. Individuals with a history of hepatitis C virus (HCV) infection must have been treated and cured. Individuals with HCV infection who are currently on treatment could be eligible if HCV viral load is undetectable.
12. Individuals with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression for at least 4 weeks. Participants need to be without requirement for steroid treatment for at least 14 days prior to the first dose of study intervention. A participant with one or two lesions that have been definitely treated with resection or focal radiation and has no symptoms is eligible after 2 weeks.
13. Based on findings from human data and/or animal studies, and their mechanisms of action, ASTX727 and olaparib can cause fetal harm when administered to a pregnant woman. For this reason, females of child-bearing potential (defined below) must agree to use adequate contraception including hormonal or barrier methods or strict abstinence for the duration of study treatment and for 6 months after last administration of study treatment. Males (with female partners of reproductive potential or who are pregnant) treated or enrolled on this protocol also must agree to use adequate contraception for the duration of study treatment, and for 3 months after last administration of study treatment. Should an individual participating in this study (or the partner of an individual participating in the study) become pregnant or suspect pregnancy, they should inform the treating physician immediately. A female is considered to be of childbearing potential (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice), unless it is documented that the individual meets either of the following two criteria: (1) has reached a postmenopausal state (>= 12 continuous months of amenorrhea with no identified cause other than menopause); or (2) has undergone surgical sterilization (i.e., hysterectomy and/or bilateral oophorectomy for removal of uterus and/or ovaries).
14. Individuals with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.

Note: Diagnosis of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML) are excluded per Exclusion # 7.

Exclusion Criteria:

1. Has received systemic anticancer therapies within 3 weeks of first dose, radiation within 2 weeks, antibody therapy within 4 weeks. Concomitant administration of Luteinizing hormone-releasing hormone (LHRH) analogues for prostate cancer and somatostatin analogues for neuroendocrine tumors are allowed as per standard of care.
2. Has not recovered from adverse events due to prior anti-cancer therapy to <= grade 1 (CTCAE v5.0) or baseline (other than alopecia).
3. Receipt of any other investigational agents or devices within 3 weeks prior to initiation of trial therapy.
4. Unable to swallow oral medications
5. Individuals who are breast-feeding/chest-feeding (because of the potential for serious adverse reactions in breastfeed infants from olaparib and ASTX727). Study participants who are lactating must agree to discontinue breast-feeding/chest-feeding for the duration of study treatment and for 1 month after the final dose of trial therapy.
6. Individuals who are pregnant (because of the potential for olaparib and ASTX727 to cause serious adverse reactions to the unborn child). Females of childbearing potential (defined below) must have a negative urine or serum pregnancy test within 72 hours prior to first administration of study drug. A female is considered to be of childbearing potential (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice), unless it is documented that the individual meets either of the following two criteria: (1) has reached a postmenopausal state (>= 12 continuous months of amenorrhea with no identified cause other than menopause); or (2) has undergone surgical sterilization (i.e., hysterectomy and/or bilateral oophorectomy for removal of uterus and/or ovaries). Individuals with any condition or social circumstance that, in the opinion of the investigator, would impair the participant's ability to comply with study activities, interfere with participant safety, or study endpoints.
7. Diagnosis of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML).
8. Taking a prohibited medication that cannot be safely discontinued or substituted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-02-07 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with treatment-emergent Adverse Events (AEs) (Phase 1 Only) | Up to 2 years
  Adverse events will be classified and graded by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0 and reported by dose level.
Percentages of dose-limiting toxicities (DLTs) (Phase 1 Only) | Up to 1 cycle (1 cycle is 28 days)
  A dose-limiting toxicity (DLT) is defined as any of the following events that are considered by the investigator to be at least possibly related to olaparib or ASTX727 and are observed during cycle 1. The percentage of participants with DLTs will be reported.
Maximum Tolerated Dose (MTD) (Phase 1 Only) | Up to 1 cycle (1 cycle is 28 days)
  The MTD is defined as the highest dose at which no more than one instance of dose-limiting toxicity (DLT) is observed among the first 6 participants treated.
Recommended Phase 2 Dose (RP2D) (Phase 1 Only) | Up to 1 cycle (1 cycle is 28 days)
  The RP2D for a planned Phase 2 trial will be selected based on the evaluation of dose-limiting toxicities and adverse events measured using CTCAE v5.0.

SECONDARY OUTCOMES:
Objective response rate (ORR) (Phase 2 only) | Up to 2 years
  ORR is defined as the proportion of participants who achieve a best overall response of confirmed complete response (CR) or confirmed partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 comparted to all participants receiving at least 1 dose of the study drug. Complete Response (CR) is defined as the disappearance of all target lesions, determined by two separate observations conducted not less than 4 weeks apart with any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm (the sum may not be "0" if there are target nodes) and there can be no appearance of new lesions. Partial response is defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD with no appearance of new lesions. Proportion and exact 90% confidence intervals will be reported.
Median Duration of overall Response (DoR) (Phase 2 only) | Up to 2 years
  DoR is defined as the duration of time from when measurement criteria are met for CR or PR (whichever is first recorded) until the date that recurrent or progressive disease (PD) is objectively documented. Median time of response with 90% confidence intervals will be summarized using the Kaplan Meier methods.
Median Duration of Stable Disease (SD) (Phase 2 only) | Up to 2 years
  Duration of SD is defined as the duration of time from start of treatment until the date that recurrent or progressive disease (PD) is objectively documented. Median duration of SD with 90% confidence intervals will be summarized using the Kaplan Meier methods.
Median Progression-Free Survival (PFS) (Phase 2 only) | Up to 2 years
  PFS is defined as duration of time from start of treatment to time of disease recurrence, progression (PD) or death from any cause, whichever occurs first. The median PFS and 90% confidence intervals will be reported using Kaplan Meier methods.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Munster, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No